CLINICAL TRIAL: NCT02055781
Title: A Randomized Controlled Phase 3 Study of Oral Pacritinib Versus Best Available Therapy in Patients With Thrombocytopenia and Primary Myelofibrosis, Post-Polycythemia Vera Myelofibrosis, or Post-Essential Thrombocythemia Myelofibrosis
Brief Title: Pacritinib Versus Best Available Therapy to Treat Patients With Myelofibrosis and Thrombocytopenia
Acronym: PAC326
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PERSIST-2 (PAC326)
Record Dates: First submitted 2014-02-03; First posted 2014-02-05 (Estimated); Results first posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-10

CONDITIONS: Primary Myelofibrosis; Post-polycythemia Vera Myelofibrosis; Post-essential Thrombocythemia Myelofibrosis
Keywords: Myelofibrosis; Post-Polycythemia Vera Myelofibrosis; Post-Essential Thrombocythemia Myelofibrosis; Primary Myelofibrosis; Polycythemia Vera; Essential Thrombocythemia; Bone Marrow Disease; Hematologic Diseases; Hemorrhagic Disorders; Splenomegaly; Pacritinib; MPN-SAF; MPN-SAF TSS; Anemia; Myeloproliferative Neoplasm; Spleen volume; Thrombocytopenia; SB1518
MeSH Terms: conditions — Primary Myelofibrosis; Polycythemia Vera; Thrombocythemia, Essential; Bone Marrow Diseases; Hematologic Diseases; Hemorrhagic Disorders; Splenomegaly; Anemia; Myeloproliferative Disorders; Thrombocytopenia | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pacritinib, Once Daily (Experimental): Pacritinib 400 mg QD
  Interventions: Drug: Pacritinib
- Pacritinib, Twice Daily (Experimental): Pacritinib 200 mg BID
  Interventions: Drug: Pacritinib
- Best Available Therapy (Active Comparator): BAT includes any physician-selected treatment for myelofibrosis, such as approved JAK2 inhibitors administered according to package insert for patients with thrombocytopenia, and may include any treatment received before study entry.
  Interventions: Drug: Best Available Therapy

INTERVENTIONS:
Drug: Pacritinib
  Arms: Pacritinib, Once Daily; Pacritinib, Twice Daily
Drug: Best Available Therapy
  Arms: Best Available Therapy

SUMMARY:
Phase 3, randomized, controlled study to evaluate the safety and efficacy of oral pacritinib compared to Best Available Therapy (BAT) in patients with thrombocytopenia and primary or secondary myelofibrosis.

DETAILED DESCRIPTION:
Multicenter, randomized, controlled, phase 3 trial comparing the safety and efficacy of pacritinib with that of BAT in patients with thrombocytopenia and primary or secondary myelofibrosis. Approximately 300 eligible patients will be randomized in a 1:1:1 allocation to pacritinib 400 mg dosed QD, pacritinib 200 mg dosed BID, or BAT (includes any physician-selected treatment for myelofibrosis, such as approved JAK2 inhibitors administered according to package insert for patients with thrombocytopenia, and may include any treatment received before study entry). Spleen volume will be measured by MRI or CT at baseline and every 12 weeks thereafter. An independent radiology facility (IRF), blind to treatment assignments, will measure spleen volumes. Patients will also be followed for safety, Leukemia Free Survival (LFS), Overall Survival (OS), frequency of red blood cell (RBC) and platelet transfusions, and other exploratory endpoints. An Independent Data Monitoring Committee (IDMC) will evaluate the safety of pacritinib.

ELIGIBILITY:
Inclusion Criteria:

* Intermediate -1 or -2 or high-risk Myelofibrosis (per Passamonti et al 2010)
* Thrombocytopenia (platelet count ≤ 100,000/µL) at any time after signing informed consent
* Palpable splenomegaly ≥ 5 cm on physical examination
* Total Symptom Score ≥ 13 on the MPN-SAF TSS 2.0, not including the inactivity question
* Patients who are platelet or red blood cell transfusion-dependent are eligible
* Adequate white blood cell counts (with low blast counts), liver function, and renal function
* At least 6 months from prior splenic irradiation
* At least 1-4 weeks since prior myelofibrosis therapy, including any erythropoietic or thrombopoietic agent
* Not pregnant, not lactating, and agree to use effective birth control
* Able and willing to undergo frequent MRI or CT assessments and complete symptom assessments using a patient-reported outcome instrument

Exclusion Criteria:

* Prior treatment with more than 2 JAK2 inhibitors or with pacritinib
* There is no maximum cumulative prior JAK2 inhibitor treatment
* History of (or plans to undergo) spleen removal surgery or allogeneic stem cell transplant
* Ongoing gastrointestinal medical condition such as Crohn's disease, Inflammatory bowel disease, chronic diarrhea, or constipation
* Active bleeding that requires hospitalization during the screening period
* Cardiovascular disease, including recent history or currently clinically symptomatic and uncontrolled: congestive heart failure, arrhythmia, angina, QTc prolongation or other QTc risk factors, myocardial infarction
* Other malignancy within last 3 years other than certain limited skin, cervical, prostate, breast, or bladder cancers
* Other ongoing, uncontrolled illnesses (including HIV infection and active hepatitis A, B, or C), psychiatric disorder, or social situation that would prevent good care on this study
* Life expectancy < 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simran Singh, Study Director — Sr. Director, Head of Clinical Operations
Locations (122):
- United States (50):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Arizona Clinical Research Center, Tucson, Arizona
  - City of Hope, Duarte, California
  - Moores Cancer Centre, La Jolla, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Stanford Cancer Center, Stanford, California
  - Rocky Mountain Cancer Center, Boulder, Colorado
  - George Washington University- Medical Faculty Associates, Washington D.C., District of Columbia
  - SCRI- Florida Cancer Specialists South Region, Fort Myers, Florida
  - SCRI - Florida Cancer Specialists North Region, St. Petersburg, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Indiana University Goshen Cancer Centre, Goshen, Indiana
  - Investigative Clinical Research of Indiana, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Siouxland Hematology-Oncology Associates, L.L.P (SHOA), Sioux City, Iowa
  - Norton Cancer Institute, Suburban, Louisville, Kentucky
  - St Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Providence Cancer Institute, Southfield, Michigan
  - Washington University School of Medicine Division of Oncology, St Louis, Missouri
  - Nebraska Hematology-Oncology, P.C., Lincoln, Nebraska
  - Hackensack University, Hackensack, New Jersey
  - Hematology-Oncology Associates of Northern Jersey, Morristown, New Jersey
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - SCRI-Oncology Hematology Care, Cincinnati, Ohio
  - Cleveland Clinic-Taussig Cancer Center, Cleveland, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Upstate Oncology Associates, Greenville, South Carolina
  - Sarah Cannon Research Institute (SCRI), Nashville, Tennessee
  - Texas Onocolgy-Baylor Sammons Cancer Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - UTMB Galveston, Galveston, Texas
  - Houston Methodist, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Huntsman Cancer Hospital, Salt Lake City, Utah
  - Virginia Cancer Specialists, Leesburg, Virginia
  - Providence Regional Cancer Partnership, Everett, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Green Bay Oncology, Green Bay, Wisconsin
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (7):
  - St George Hospital, Kogarah, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Health - Monash Medical Centre, Clayton, Victoria
  - Perth Blood Institute, Nedlands, Western Australia
  - Haematology and Oncology Clinics of Australia, Chermside
  - Prince of Wales Hospital, Randwick
- Belgium (7):
  - Centre Hospitalier de Jolimont-Lobbes, Haine-Saint-Paul, Hainaut
  - ZNA - Stuivenberg, Antwerp
  - AZ Sint Jan Brugge-Oostende AV, Bruges
  - Hopital Brugmann, Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - St Augustinus, Wilrijk
  - UC Louvain, Yvoir
- Canada (2):
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Princess Margaret Cancer Center, Toronto, Ontario
- Czechia (4):
  - Fakultní nemocnice Brno, Brno, NAP
  - Faculty Hospital Olomouc, Olomouc, NAP
  - Fakultní nemocnice Plzeň, Pilsen, NAP
  - University Hospital Hradec Kralove, Králová
- France (12):
  - Chu d'Amiens Hopital Sud, Amiens, Cedex 1
  - Hôpital Caremeau, Nîmes, Cedex 9
  - CHU Rennes, Rennes, Cedex 9
  - CHU Purpan, Toulouse, Cedex 9
  - CH de Mulhouse, Mulhouse, Cedex
  - CHU de CAEN, Caen
  - Centre Hospitalier de Lens, Lens
  - Hopital l'Archet, CHU de Nice, Nice
  - Saint Antoine Hospital, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Strasbourg, Strasbourg
  - Institut Gustave Roussy, Villejuif
- Germany (10):
  - Charite-Medical University, Berlin
  - Klinik I fur Innere Medizin, Universitat Koln, Cologne
  - Gemeinschaftspraxis Hämatologie/Onkologie, Dresden
  - University Hospital Essen, Essen
  - Uniklinik Freiburg, Freiburg im Breisgau
  - Universitatsklinikum Halle (Saale), Halle
  - University Hospital Leipzig, Leipzig
  - Städtisches Klinikum München GmbH, München
  - University of Munster, Münster
  - University Hospital Ulm, Ulm
- Hungary (6):
  - Semmelweis Egyetem AOK, Budapest
  - University of Debrecen, Belgyogyaszati Intezet, Debrecen
  - Bekes Megyei Pandy Kalman Korhaz, Gyula
  - Kaposi Mór Oktató Kórház, Kaposvár
  - SZTE II. sz Belgyogyoszati Klinika es Kardiologiai Kozpont, Szeged
  - Jász-Nagykun-Szolnok Megyei Hetényi Géza Kórház-Rendelőint, Szolnok
- Netherlands (2):
  - University Hospital Maastricht, Maastricht
  - Erasmus MC, Rotterdam
- New Zealand (5):
  - Auckland District Health Board, Auckland City Hospital, Auckland
  - Middlemore Hospital, Auckland
  - Canterbury District Health Board, Christchurch
  - North Shore Hospital, Takapuna
  - CCDHB - Wellington Hospital, Wellington
- Russia (7):
  - Bashkir State Medical University, Ufa, Bashkortostan Republic
  - Saratov State Medical University, Saratov, Saratov Oblast
  - National Haematology Research Center, Moscow
  - Republican Hopsital n.a. V.A. Baranov, Petrozavodsk
  - Ryazan Regional Clinical Hospital, Ryazan
  - Russian Research Institute of Hematology and Transfusiology, Saint Petersburg
  - Military Medical Academy n.a. S.M. Kirov, Saint Petersburg
- United Kingdom (10):
  - Royal Liverpool University Hospital, Liverpool, Merseyside
  - Belfast Health and Social Care Trust, Belfast, Northern Ireland
  - Birmingham Heartlands Hospital, Birmingham
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Leicester Royal Infirmary, Leicester
  - Guy's Hospital, London
  - Hammersmith Hosp - ICH NHS Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Oxford University Hospitals NHS Trust, Oxford
  - Royal Hallamshire Hospital, Sheffield

REFERENCES:
- [Background] Mascarenhas J, Hoffman R, Talpaz M, Gerds AT, Stein B, Gupta V, Szoke A, Drummond M, Pristupa A, Granston T, Daly R, Al-Fayoumi S, Callahan JA, Singer JW, Gotlib J, Jamieson C, Harrison C, Mesa R, Verstovsek S. Pacritinib vs Best Available Therapy, Including Ruxolitinib, in Patients With Myelofibrosis: A Randomized Clinical Trial. JAMA Oncol. 2018 May 1;4(5):652-659. doi: 10.1001/jamaoncol.2017.5818. PMID 29522138
- [Derived] Ajufo H, Bewersdorf JP, Harrison C, Palandri F, Mascarenhas J, Palmer J, Gerds A, Kiladjian JJ, Buckley S, Derkach A, Roman-Torres K, Rampal RK. Pacritinib Response Is Associated With Overall Survival in Myelofibrosis: PERSIST-2 Landmark Analysis of Survival. Eur J Haematol. 2025 Feb;114(2):238-247. doi: 10.1111/ejh.14321. Epub 2024 Oct 14. PMID 39400386
- [Derived] Verstovsek S, Mesa R, Talpaz M, Kiladjian JJ, Harrison CN, Oh ST, Vannucchi AM, Rampal R, Scott BL, Buckley SA, Craig AR, Roman-Torres K, Mascarenhas JO. Retrospective analysis of pacritinib in patients with myelofibrosis and severe thrombocytopenia. Haematologica. 2022 Jul 1;107(7):1599-1607. doi: 10.3324/haematol.2021.279415. PMID 34551507
- [Derived] Tremblay D, Mesa R, Scott B, Buckley S, Roman-Torres K, Verstovsek S, Mascarenhas J. Pacritinib demonstrates spleen volume reduction in patients with myelofibrosis independent of JAK2V617F allele burden. Blood Adv. 2020 Dec 8;4(23):5929-5935. doi: 10.1182/bloodadvances.2020002970. PMID 33275766

RESULTS

PARTICIPANT FLOW:
Groups:
- Pacritinib, QD: Pacritinib 400 mg QD
- Pacritinib, BID: Pacritinib 200 mg BID
Period: Overall Study
Arm/Group | Pacritinib, QD | Pacritinib, BID | Best Available Therapy
Started | 104 | 107 | 100
Completed | 62 | 79 | 63
Not Completed | 42 | 28 | 37

BASELINE CHARACTERISTICS:
Population: Represents Intent To Treat population (number of randomized patients)
Groups:
- Pacritinib, Once Daily: Pacritinib 400 mg, once daily
- Pacritinib, Twice Daily: Pacritinib 200 mg, twice daily
- Total: Total of all reporting groups
Arm/Group | Pacritinib, Once Daily | Pacritinib, Twice Daily | Best Available Therapy | Total
Number analyzed (Participants) | 104 | 107 | 100 | 311
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 32 | 41 | 32 | 105
  Between 18 and 65 years | 70 | 65 | 68 | 203
  >=65 years | 2 | 1 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (8.55) | 65.9 (8.75) | 66.9 (9.75) | 67.2 (9.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 44 | 45 | 140
  Male | 53 | 63 | 55 | 171
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 4 | 6 | 3 | 13
  Canada | 5 | 2 | 4 | 11
  Netherlands | 0 | 1 | 1 | 2
  Belgium | 2 | 2 | 1 | 5
  Hungary | 9 | 8 | 7 | 24
  United States | 44 | 44 | 43 | 131
  Czechia | 2 | 4 | 5 | 11
  United Kingdom | 5 | 11 | 11 | 27
  Australia | 4 | 5 | 4 | 13
  France | 8 | 10 | 9 | 27
  Germany | 10 | 4 | 3 | 17
  Russia | 11 | 10 | 9 | 30

OUTCOME MEASURES:

1. Primary Outcome: Spleen Volume Reduction
Description: Proportion of patients achieving a ≥ 35% reduction in spleen volume from baseline to week 24 as measured by magnetic resonance imaging (MRI) or computed tomography (CT).
Time Frame: Baseline to Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Pacritinib, Once Daily | Pacritinib, Twice Daily | Best Available Therapy
Number analyzed (Participants) | 75 | 74 | 72
Participants | 11 | 16 | 2
Statistical Analysis 1: Comparison: Pacritinib, Once Daily vs Pacritinib, Twice Daily vs Best Available Therapy; BAT arm compared to pooled pacritinib arms (QD + BID - ITT Efficacy); Test type: Superiority; p = 0.0011, Fisher Exact
Statistical Analysis 2: Comparison: Pacritinib, Once Daily vs Best Available Therapy; Test type: Superiority; p = 0.0173, Fisher Exact
Statistical Analysis 3: Comparison: Pacritinib, Twice Daily vs Best Available Therapy; Test type: Superiority; p = 0.0007, Fisher Exact

2. Primary Outcome: Total Symptom Score (TSS) Reduction
Description: Proportion of patients achieving a ≥ 50% reduction in the total symptom score from baseline to Week 24 on the Myeloproliferative Neoplasm Symptom Assessment Form 2.0 (MPN-SAF TSS 2.0). Responses (on a scale from 0 [absent] to 10 [worst imaginable]) to questions about symptoms (tiredness, early satiety, abdominal discomfort, night sweats, pruritus, bone pain, and pain under the ribs on the left side) were used to calculate the TSS.
Time Frame: Baseline to Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Pacritinib, Once Daily | Pacritinib, Twice Daily | Best Available Therapy
Number analyzed (Participants) | 75 | 74 | 72
Participants | 13 | 24 | 10
Statistical Analysis 1: Comparison: Pacritinib, Once Daily vs Pacritinib, Twice Daily vs Best Available Therapy; BAT arm compared to pooled pacritinib arms (QD + BID - ITT Efficacy); Test type: Superiority; p = 0.0791, Fisher Exact
Statistical Analysis 2: Comparison: Pacritinib, Once Daily vs Best Available Therapy; Test type: Superiority; p = 0.6524, Fisher Exact
Statistical Analysis 3: Comparison: Pacritinib, Twice Daily vs Best Available Therapy; Test type: Superiority; p = 0.0106, Fisher Exact

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent through 30 days after the last study treatment.
Description: All-Cause Mortality was assessed in the Total Randomized Population (n=311). Serious Adverse Events and Other (Not Including Serious) Adverse Events were assessed in the Safety Population (n=308).
Arm/Group | Pacritinib, Once Daily | Pacritinib, Twice Daily | Best Available Therapy
All-Cause Mortality (participants affected / at risk) | 22/104 | 20/107 | 20/100
Serious Adverse Events (participants affected / at risk) | 48/104 | 50/106 | 30/98
Other Adverse Events (participants affected / at risk) | 104/104 | 100/106 | 87/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pacritinib, Once Daily (N=104) | Pacritinib, Twice Daily (N=106) | Best Available Therapy (N=98)
Deep vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 4 (4) | 3 (3) | 3 (3)
Pyrexia (General disorders) | 2 (2) | 3 (3) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 4 (4) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 0 (0) | 3 (3)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 8 (8) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 6 (6) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Haemorrholdal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 5 (5) | 2 (2) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Periarthrtis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 6 (6) | 4 (4)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphocytic infiltration (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tooth socket haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hodgkin's disease nodular sclerosis stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Central nervous system lesion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Encephalomalacia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Intracranial venous sinus thrombosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Meningorrhagia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder perforation (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ovarian rupture (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Neurological decompensation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pacritinib, Once Daily (N=104) | Pacritinib, Twice Daily (N=106) | Best Available Therapy (N=98)
Contusion (Injury, poisoning and procedural complications) | 7 (7) | 10 (10) | 8 (8)
Fall (Injury, poisoning and procedural complications) | 7 (7) | 5 (5) | 3 (3)
Weight decreased (Investigations) | 4 (4) | 7 (7) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 13 (13) | 13 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 9 (9) | 10 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 11 (11) | 9 (9)
Thrombocytopenia (Blood and lymphatic system disorders) | 34 (34) | 36 (36) | 23 (23)
Anaemia (Blood and lymphatic system disorders) | 29 | 25 | 15 (15)
Neutropenia (Blood and lymphatic system disorders) | 9 (9) | 9 (9) | 6 (6)
Dizziness (Nervous system disorders) | 15 (15) | 16 (16) | 5 (5)
Dysgeusia (Nervous system disorders) | 8 (8) | 8 (8) | 0 (0)
Headache (Nervous system disorders) | 6 (6) | 9 (9) | 5 (5)
Fatigue (General disorders) | 18 (18) | 18 (18) | 16 (16)
Oedema peripheral (General disorders) | 14 (14) | 21 (21) | 15 (15)
Asthenia (General disorders) | 5 (5) | 3 (3) | 6 (6)
Early satiety (General disorders) | 1 (1) | 3 (3) | 5 (5)
Pyrexia (General disorders) | 11 (11) | 16 (16) | 3 (3)
Insomnia (Psychiatric disorders) | 12 (12) | 10 (10) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 70 (70) | 51 (51) | 15 (15)
Nausea (Gastrointestinal disorders) | 39 (39) | 34 (34) | 11 (11)
Vomiting (Gastrointestinal disorders) | 22 (22) | 20 (20) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 20 (20) | 10 (10) | 19 (19)
Abdmonial distension (Gastrointestinal disorders) | 3 (3) | 6 (6) | 6 (6)
Abdominal pain upper (Gastrointestinal disorders) | 6 (6) | 6 (6) | 6 (6)
Constipation (Gastrointestinal disorders) | 15 (15) | 8 (8) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (10) | 11 (11) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 8 (8) | 5 (5)
Night sweats (Skin and subcutaneous tissue disorders) | 8 (8) | 8 (8) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 9 (9) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 7 (7) | 7 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7) | 10 (10) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 13 (13) | 13 (13) | 11 (11)
Upper respiratory tract infection (Infections and infestations) | 8 (8) | 11 (11) | 6 (6)
Conjunctival haemorrhage (Eye disorders) | 3 (3) | 6 (6) | 4 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (6) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 8 (8) | 9 (9) | 4 (4)
Urinary tract infection (Infections and infestations) | 8 (8) | 4 (4) | 2 (2)
Bronchitis (Infections and infestations) | 3 (3) | 6 (6) | 3 (3)
Electrocardiogram QT prolonged (Investigations) | 6 (6) | 2 (2) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 6 (6) | 3 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (7) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 6 (6) | 3 (3) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1) | 2 (2)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (7) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (6) | 0 (0)
Haematoma (Vascular disorders) | 3 (3) | 6 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other